CLINICAL TRIAL: NCT03676556
Title: Double-blind Randomized Clinical Trial to Evaluate the Reduction of Pain in the Wounds Treatment Previously Applying Lidocaine Topical Solution vs Placebo, in the Outpatients Area.
Brief Title: To Evaluate Reduction of Pain in Wounds Treatment Previously Applying Lidocaine Topical Solution vs Placebo.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Ana Sanchez Allueva, Anesthesiologist, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LIDO2017
Record Dates: First submitted 2018-03-26; First posted 2018-09-18 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Wound; Anesthesia, Local
Keywords: wound treatment; lidocaine; pain reduction; local anesthetic
MeSH Terms: conditions — Wounds and Injuries | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical lidocaine (Active Comparator): 23 patients will recieve lidocaine solution before wound treatment
  Interventions: Drug: Lidocaine
- Saline serum (Placebo Comparator): 23 patients will recieve saline solution before wound treatment
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Lidocaine — Two sterile gauzes will be dampen with the content of the syringe (20ml lidocaine 0.5%) and apply on the wound. After 7-15minutes of waiting to the effect, the wound treatment will start.
  Arms: Topical lidocaine
Drug: Saline Solution — Two sterile gauzes will be dampen with the content of the syringe (20ml saline serum) and apply on the wound. After 7-15minutes of waiting to the effect, the wound treatment will start.
  Arms: Saline serum

SUMMARY:
The purpose of this study is to evaluate if applying a lidocaine topical solution before wounds treatment decreases the pain of the procedure in comparison with placebo solution.

DETAILED DESCRIPTION:
The manipulation of the wounds for its treatment is a painful process and there is currently no marketed any topical drug to decrease this suffering.

The objective of this study is to demonstrate that lidocaine topical solution applied prior to wounds treatment, reduces the pain of the procedure compared to the treatment done after application of placebo solution. In addition, if the process was less painful, the consumption of systemic analgesics would be reduced (or eliminated) and, therefore, also its secondary effects.

It is a single-center clinical trial, prospective, randomised, double-blind, placebo-controlled study that will include 46 patients (23 lidocaine group, 23 placebo group) who presents painful wounds during treatment in the Bellvitge University Hospital (HUB) outpatients area.

The Pharmaceutical Department of HUB prepares a dilution of lidocaine 0.5% in 20ml disposable syringes and identical disposable syringes containing 20ml saline solution (process authorized by the Spanish Agency of Medicines and Sanitary Products).

When a patient arrives at the outpatient area (dermatology or plastic surgery departments) to treat a wound, the nursery or the doctor who does the procedure evaluates the pain during the treatment. If it is 5 or more points according the "Verbal Numerical Scale" (VNS), the nursery will explain to the patient the possibility of being a participant in this study, and give the information document. If the patient is interested, the doctor of the Pain Department will be warned and an EKG and a pregnancy test (if the patient is a woman in fertile age) will be done.

The doctor of the Pain Department will answer to any question about the study, will collect the medical record, will evaluate de EKG and the pregnancy test if it was done. Counting with all this information, and checking inclusion/exclusion criterias, the patient will be recluted. The patient will be ask to register in a data document any analgesic needed in the following 24 hours and also to register the VNS punctuation (0-10) 24 hours after the procedure, and to bring all this information the day of the next wound treatment. To avoid bias, the doctor of the Pain Department, will ask the patient to take the same analgesics the day of the study.

Between the basal wound treatment (it is, the day of the recruitment) and the wound treatment of the study (it will be the next wound treatment, when lidocaine or placebo will be applied, depending on the random list) there will not elapse more than 10 days.

The random process, will be done in the Pharmaceutical Department, following a table of random, starting at numer 01. The pair number will receive lidocaine, and the odd numbers saline solution. Each syringe will be named by an ordinary number, according with the recruitment number. And they will give this syringes to the outpatient area.

The day of the study, the nursery or the Pain Department doctor will record the VNS punctuation before treatment; then the nursery will apply wetted gauzes with the study solution and will wait 7-15 minutes to effect (exactly time counted and registrered with a chronometer). After this time the habitual treatment will be applied and at this moment the pain in the VNS will be recored. The nursery or the Pain Department doctor will be attentive to any secondary effect appears. And finally, the nursery will ask again about the pain 15 minutes after the procedure.

The nursery or the Pain Department doctor will ask to the patient to record the analgesics need in the following 24 hours and, after this period, the Pain Department doctor will call the patient to ask about this record, about the pain at 24 hours after the procedure and if any secondary effect has been detected.

Comparing the procedures carried out after lidocaine solution with saline solution, the investigators will evaluate the reduction of pain in the wounds treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has accepted and signed the informed consent before the random process.
* Women or men aged more than 18 years
* Patients with painful wound treatments (> or = 5) who come to outgoing area for the treatment
* Wounds or sores of any aetiology sauf arterial deficit that implies at minimum dermis or epidermis, it is, II to IV degree in the Spanish Classification of Sores made by the "National Group to Study and Management of Pressure Ulcers and Chronic Wounds" (GNEAUPP).
* Women in fertile age with pregnancy test negative

Exclusion Criteria:

* Precedents of allergic reaction to local anesthesics type amides.
* Wounds or sores degree I on the GNEAUPP Classification (it is, without discontinuity of skin).
* Wounds or sores too large (which requirej more than 40 ml of solution to cover)
* Wounds around the eyes
* Wounds secondary to arterial deficit
* Patients who presents disturbance of cardiac conduction: atrioventricular block (second or third degree) or bifascicular block
* Patients with altered level of consciousness (Glasgow Coma Scale value less than 14)
* Patients following hemodialysis, peritoneal dialysis or continuous hemofiltration treatment
* Patients suffering moderate or severe hepatic insufficiency
* Pregnant or lactating women
* Once the patient has already participate in the study during a previous wound treatment
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Register the VNS (Verbal Numeric Scale) punctuation (between 0 it is not pain, and 10 it is unbearable pain) during wound treatment. | Maximum 10 days between the day of the recruitement and the treatment of the study.
  We will register the VNS punctuation during the wound treatment the day of the recruitment and also the day of study. We expect to obtain less punctuation when lidocaine solution has been administrated vs saline solution.

SECONDARY OUTCOMES:
Register the VNS (Verbal Numeric Scale) punctuation (between 0 it is not pain, and 10 it is unbearable pain)15 minutes after wound treatment has finished. | 15 minutes after each wound treatment of the study has finished.
  We will register the VNS punctuation 15 minutes after wound treatment has finished, the day of the recruitment and also the day of study. We expect to obtain less punctuation when lidocaine solution has been administrated vs saline solution.
Register the VNS (Verbal Numeric Scale) punctuation (between 0 it is not pain, and 10 it is unbearable pain) at 24 hours after each wound treatment of the study. | At 24 hours after each wound treatment of the study
  We will give to the patient a data document to register the VNS punctuation at 24 hours after each wound treatment of the study.
  t the day of recruitment. The patient will give to the nursery this data document the day of the study treatment. 24 hours after the study treatment, the Pain Department doctor will call to the patient by phone, to get the same information than in the data document. We expect to obtain less VNS punctuation when lidocaine solution has been administrated vs saline solution.
Register if appears any side effect: local (alterations in the skin, pruritus...) or systemic (tinnitus, metallic flavor, arrhythmia...) during each procedure and in the next 24 hours after each wound treatment. | Up to 24 hours after each wound treatment of the study
  Registering if any side effect (local or systemic) appears during each procedure and in the next 24 hours after each wound treatment.
Register the exact time to application of the wet gauzes with the study solution (between 7 and 15 minutes) | Between 7 and 15 minutes
  The nursery will record the time of application of the wet gauzes with a chronometer. This time of application has to be always between 7 and 15 minutes.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Ana Sánchez Allueva, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona

IPD SHARING:
Plan to Share IPD: No
We do not give information to any other people

REFERENCES:
- [Background] Ozgocmen S, Kaya A, Coskun BK. Topical lidocaine helps reduce pain of digital ulcers in systemic sclerosis (scleroderma). Clin Rheumatol. 2006 May;25(3):378-9. doi: 10.1007/s10067-005-0016-1. Epub 2005 Oct 7. No abstract available. PMID 16211339
- [Background] Franz-Montan M, Ranali J, Ramacciato JC, de Andrade ED, Volpato MC, Groppo FC. Ulceration of gingival mucosa after topical application of EMLA: report of four cases. Br Dent J. 2008 Feb 9;204(3):133-4. doi: 10.1038/bdj.2008.48. PMID 18264061
- [Background] Stahl M, Meyer C, Haas E, Glaenz T, Zutt M. Leg ulcer progression caused by topical anesthesia with EMLA cream. J Dtsch Dermatol Ges. 2008 Jul;6(7):566-8. doi: 10.1111/j.1610-0387.2007.06532.x. Epub 2007 Oct 17. English, German. PMID 17941883
- [Background] Boulinguez S, Sparsa A, Bouyssou-Gauthier ML, Bedane C, Bonnetblanc JM. Adverse effects associated with EMLA cream used as topical anesthetic for the mechanical debridement of leg ulcers. J Am Acad Dermatol. 2000 Jan;42(1 Pt 1):146-8. doi: 10.1016/s0190-9622(00)90030-6. No abstract available. PMID 10607341
- [Background] Yamashita S, Sato S, Kakiuchi Y, Miyabe M, Yamaguchi H. Lidocaine toxicity during frequent viscous lidocaine use for painful tongue ulcer. J Pain Symptom Manage. 2002 Nov;24(5):543-5. doi: 10.1016/s0885-3924(02)00498-0. PMID 12547053
- [Background] Davis MD, Adams A. Lidocaine patch for the management of leg ulcer pain. J Am Acad Dermatol. 2006 Nov;55(5 Suppl):S126-7. doi: 10.1016/j.jaad.2006.02.056. No abstract available. PMID 17052535
- [Background] Sliti N, Zaraa I, Daoud L, Trojett S, Letaief I, Mokni M, Jeddi A, Ben Osman A. [Acute bilateral palpebral necrosis: a rare complication of local anaesthesia]. Ann Dermatol Venereol. 2010 Jan;137(1):84-5. doi: 10.1016/j.annder.2009.10.001. Epub 2009 Nov 20. No abstract available. French. PMID 20110079
- [Background] Claeys A, Gaudy-Marqueste C, Pauly V, Pelletier F, Truchetet F, Boye T, Aubin F, Schmutz JL, Grob JJ, Richard MA. Management of pain associated with debridement of leg ulcers: a randomized, multicentre, pilot study comparing nitrous oxide-oxygen mixture inhalation and lidocaine-prilocaine cream. J Eur Acad Dermatol Venereol. 2011 Feb;25(2):138-44. doi: 10.1111/j.1468-3083.2010.03720.x. Epub 2010 Jun 21. PMID 20569291
- [Background] Holst RG, Kristofferson A. Lidocaine-prilocaine cream (EMLA Cream) as a topical anaesthetic for the cleansing of leg ulcers. The effect of length of application time. Eur J Dermatol. 1998 Jun;8(4):245-7. PMID 9649697
- [Background] Lok C, Paul C, Amblard P, Bessis D, Debure C, Faivre B, Guillot B, Ortonne JP, Huledal G, Kalis B. EMLA cream as a topical anesthetic for the repeated mechanical debridement of venous leg ulcers: a double-blind, placebo-controlled study. J Am Acad Dermatol. 1999 Feb;40(2 Pt 1):208-13. doi: 10.1016/s0190-9622(99)70190-8. PMID 10025747
- [Background] Bershow A, Warshaw E. Cutaneous reactions to transdermal therapeutic systems. Dermatitis. 2011 Jul-Aug;22(4):193-203. PMID 21781635
- [Background] Briggs M, Nelson EA, Martyn-St James M. Topical agents or dressings for pain in venous leg ulcers. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD001177. doi: 10.1002/14651858.CD001177.pub3. PMID 23152206
- [Background] Brolmann FE, Ubbink DT, Nelson EA, Munte K, van der Horst CM, Vermeulen H. Evidence-based decisions for local and systemic wound care. Br J Surg. 2012 Sep;99(9):1172-83. doi: 10.1002/bjs.8810. Epub 2012 Jul 6. PMID 22777856
- [Background] Cooper SM, Hofman D, Burge SM. Leg ulcers and pain: a review. Int J Low Extrem Wounds. 2003 Dec;2(4):189-97. doi: 10.1177/1534734603260556. PMID 15866847
- [Background] Sobanko JF, Miller CJ, Alster TS. Topical anesthetics for dermatologic procedures: a review. Dermatol Surg. 2012 May;38(5):709-21. doi: 10.1111/j.1524-4725.2011.02271.x. Epub 2012 Jan 13. PMID 22243434
- [Background] Descroix V, Coudert AE, Vige A, Durand JP, Toupenay S, Molla M, Pompignoli M, Missika P, Allaert FA. Efficacy of topical 1% lidocaine in the symptomatic treatment of pain associated with oral mucosal trauma or minor oral aphthous ulcer: a randomized, double-blind, placebo-controlled, parallel-group, single-dose study. J Orofac Pain. 2011 Fall;25(4):327-32. PMID 22247928
- [Background] Vanscheidt W, Sadjadi Z, Lillieborg S. EMLA anaesthetic cream for sharp leg ulcer debridement: a review of the clinical evidence for analgesic efficacy and tolerability. Eur J Dermatol. 2001 Mar-Apr;11(2):90-6. PMID 11275800